CLINICAL TRIAL: NCT03687606
Title: Efficacy and Safety of Long Term Use of hCG or hCG Plus hMG in the Treatment of Male Patients With Isolated Hypogonadotropic Hypogonadism: an Open, Randomized Controlled Study
Brief Title: Efficacy and Safety of Long Term Use of hCG or hCG Plus hMG in Males With Isolated Hypogonadotropic Hypogonadism (IHH)
Acronym: IHH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jihong Liu, Principal Investigator, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20180906
Record Dates: First submitted 2018-09-16; First posted 2018-09-27 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Isolated Hypogonadotropic Hypogonadism; Kallmann Syndrome; Infertility
Keywords: Gonadotropin treatment; human chorionic gonadotropin; human menopausal gonadotropin
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome; Infertility | interventions — Chorionic Gonadotropin; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Human Chorionic Gonadotropin alone (Active Comparator): Human Chorionic Gonadotropin 2000U~6000U, intramuscular injection, two times per week for 3 years.
  Interventions: Drug: Human Chorionic Gonadotropin
- hCG alone for 6 months then hMG added (Experimental): Human Chorionic Gonadotropin 2000U~6000U, intramuscular injection, two times per week for six months, then 75~150IU human menopausal gonadotropin, intramuscular injection, two times per week, was added and last for the next 30 months.
  Interventions: Drug: Human Chorionic Gonadotropin; Drug: human menopausal gonadotropin
- hCG and hMG (Experimental): Human Chorionic Gonadotropin 2000U~6000U and 75~150IU human menopausal gonadotropin, intramuscular injection, two times per week for 3 years.
  Interventions: Drug: Human Chorionic Gonadotropin; Drug: human menopausal gonadotropin

INTERVENTIONS:
Drug: Human Chorionic Gonadotropin — White freeze-dried cake or powder with specifications of 1000U, 2000U, 5000U.
  Other Names: hCG
Drug: human menopausal gonadotropin — White freeze-dried cake or powder with specification of 75IU.
  Other Names: hMG
  Arms: hCG alone for 6 months then hMG added; hCG and hMG

SUMMARY:
This study will evaluate the efficacy and safety of long term use of hCG alone or hCG plus hMG in the treatment of male patients with isolated hypogonadotropic hypogonadism (IHH). One third of the participants will receive hCG treatment alone and the other third of the participants will receive hCG treatment alone for six months, then the hMG will be added. And the last third of the participants will receive hCG and hMG treatment since the beginning of the treatment.

DETAILED DESCRIPTION:
The efficacy of hCG alone or hCG plus hMG in the treatment of male IHH patients was reported in some studies. However, these studies were mostly non-randomized controlled studies with small size of samples and short follow-up time. There was also no reported study which aimed to compare the efficacy and safety of long term use of hCG or hCG plus hMG in the treatment of male patients with IHH. So the difference in the efficacy and safety between long term use of hCG alone and hCG plus hMG in the treatment of IHH is unknown. In different reported studies, the hCG plus hMG treatment had two regimens: using hCG alone for six month, then hMG was added and using hCG plus hMG since the beginning of the treatment. The difference in the efficacy and safety between the above two regimes is also unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, ≤ 45 years old;
2. Adolescent dysplasia or loss of puberty: Genital Tanner score ﹤ 5, pubic hair Tanner score ﹤ 5;
3. Serum FSH and LH levels are low or in normal low value, testosterone was lower than normal range (1.75ng / ml, the lower limit of the normal blood testosterone reference range of Tongji Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology);
4. With or without olfactory loss/reduction;
5. Other pituitary hormone levels are normal;
6. Head MRI examination is normal;
7. Fertility is desired currently or will be desired in the future;
8. Understand and sign the informed consent form.

Exclusion Criteria:

1. Primary hypogonadism;
2. Acquired hypogonadotrophic hypogonadism;
3. A history of treatment with pulsed GnRH, hCG and FSH related hormones;
4. Receive testosterone replacement therapy for more than 6 months;
5. History of cryptorchidism or cryptorchidism;
6. The sperm density before treatment ≥1×10^6/ml;
7. Moderate or severe liver and kidney dysfunction (ALT>120IU/L, AST>80IU/L, CR>115μmol/L);
8. The karyotype is 45,X or 47,XXY and 48, XXXY and other abnormal karyotypes;
9. True hermaphroditism and pseudohermaphroditism;
10. Sex hormone abnormalities caused by adrenal lesions;
11. Hypogonadism secondary to other systemic diseases;
12. Abnormal secretion of hormones caused by brain lesions (such as pituitary tumors);
13. There are other hormone abnormalities in the pituitary;
14. There are contraindications for the treatment with hCG or hMG.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sperm density | 6 months.
  Sperm density will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.

SECONDARY OUTCOMES:
Semen volume | 6 months.
  Sperm volume will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
Sperm activity | 6 months.
  Sperm activity will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
The time for sperm to appear during treatment | 6 months.
  The time for the sperm firstly appeared in the semen will be recorded.
Serum testosterone levels | 3 months.
  The serum testosterone levels will be tested in every visit.
Testicular volume | 3 months.
  Testicular volume will be measured using a Prader orchidometer.
Penis length | 3 months.
  Penis length will be measured from the pubic symphysis to glans using a vernier caliper.
Pubic hair | 3 months.
  Pubic hair will be evaluated according to Tanner pubertal stages.
Genitalia | 3 months.
  Genitalia will be evaluated according to Tanner pubertal stages.

OTHER OUTCOMES:
Height | 3 months.
  Height will be measured at every visit.
Weight | 3 months.
  Weight will be measured at every visit.
Feeling of inferiority scale score | 3 months.
  Feeling of inferiority scale scores will be obtained using feeling of inferiority scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, M.D, Principal Investigator — Departments of Urology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China.
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available with 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the external independent review panel and Tongji hospital. Requester will be reqiured to sign a Data Acces Agreement.

REFERENCES:
- [Background] Zacharin M, Sabin MA, Nair VV, Dabadghao P. Addition of recombinant follicle-stimulating hormone to human chorionic gonadotropin treatment in adolescents and young adults with hypogonadotropic hypogonadism promotes normal testicular growth and may promote early spermatogenesis. Fertil Steril. 2012 Oct;98(4):836-42. doi: 10.1016/j.fertnstert.2012.06.022. Epub 2012 Jul 3. PMID 22763096
- [Background] Matsumoto AM, Snyder PJ, Bhasin S, Martin K, Weber T, Winters S, Spratt D, Brentzel J, O'Dea L. Stimulation of spermatogenesis with recombinant human follicle-stimulating hormone (follitropin alfa; GONAL-f): long-term treatment in azoospermic men with hypogonadotropic hypogonadism. Fertil Steril. 2009 Sep;92(3):979-990. doi: 10.1016/j.fertnstert.2008.07.1742. Epub 2008 Oct 18. PMID 18930190